CLINICAL TRIAL: NCT03555513
Title: The Frequency and Risk Factors of Delayed Graft Function in Living Donor Kidney Transplantation and Its Clinical Impact in Part of Middle East
Brief Title: The Frequency and Risk Factors of Delayed Graft Function
Status: Completed | Type: Observational
Sponsor: nooshin dalili (Other)
Responsible Party: Sponsor-Investigator, nooshin dalili, Assistant Professor of SBMU, Shahid Beheshti University of Medical Sciences
Organization: Shahid Beheshti University of Medical Sciences (Other)
Other Study IDs: SB24576H
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Last update posted 2018-06-13 (Actual); Status verified 2018-06

CONDITIONS: Delayed Graft Function; Kidney Transplant; Complications
MeSH Terms: conditions — Delayed Graft Function

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- living kidney transplanted patients: Any patients over 18 who received kidney transplantation from living donor
  Interventions: Procedure: living kidney transplantation

INTERVENTIONS:
Procedure: living kidney transplantation — receiving kidney transplantation from living donor

SUMMARY:
Delayed graft function (DGF) is an important phenomenon after kidney transplantation with direct and indirect implication on graft survival. Although its incidence and risk factors have been studied after cadaveric kidney transplantation cases, only few data is available regarding transplants from living donors. The present study was performed to investigate the frequency and risk factors of DGF among living-unrelated kidney transplant recipients among three transplant centers in part of Middle East.

DETAILED DESCRIPTION:
In this multi-center retrospective study, data from 480 transplanted patients had been collected from existing local hospital registries in three countries (Iran, Kingdom of Saudi Arabia (KSA), and Kuwait) with 3 years post transplantation follow-up. Data for this study was collected based on routine clinical practice of medical practitioners across the participating countries. A case report data collecting form was designed for gathering the data including the recipient and donor's characteristics prior to transplantation, and after transplantation up to three years post transplantation. Using binary logistic regression analysis, the potential risk factors for occurrence of DGF in living donor transplantations were tested. Graft and patient survival at 1, 2 and 3 years depending on follow-up time was evaluated.

ELIGIBILITY:
Inclusion Criteria:

Living donor kidney recipients with complete prior transplantation data and 3 years post transplantation follow up, including those who died during the observation period

Exclusion Criteria:

kidney recipients younger than 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A case report data collecting form was designed for gathering the following data: the recipients and donors characteristics prior to transplantation, time on dialysis (months), first or second transplantation, panel reactive antibody (PRA) and human leukocyte antigen (HLA) mismatch, frequency of DGF, renal function, cold and warm ischemia time, immunosuppressive regimens (induction, if any used), adverse events, acute and chronic graft rejection, graft survival and patient survival at 1, 2 and 3 years follow-up.It was planned to recruit 500 patients, from 3 centers in 3 countries of Middle east. Distribution by country or region was as following :Iran (n=300), Kuwait (n=100) and KSA (n=100) subjects . As it was a retrospective disease registry with no access or possibility to recall patients, obtaining informed consent form from patients was waived up to the local regulatory processes. Approvals were obtained from each site to access patients' records and collect their data.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
incidence of delayed graft function | 3 years

SECONDARY OUTCOMES:
risk factors of DGF | three years

CONTACTS AND LOCATIONS:
Overall Officials: Shahid Beheshti University of Medical Sciences, Medical, Principal Investigator — Shahid Beheshti University of Medical Sciences

IPD SHARING:
Plan to Share IPD: No